CLINICAL TRIAL: NCT03943602
Title: Cabozantinib in Patients With Advanced Penile Squamous Cell Carcinoma (PSCC): an Open-label, Single-center, Phase 2, Single-arm Trial (CaboPen)
Brief Title: Cabozantinib in Patients With Advanced Penile Squamous Cell Carcinoma (PSCC) (CaboPen)
Acronym: CaboPen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaboPen
Record Dates: First submitted 2019-03-26; First posted 2019-05-09 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Penile Squamous Cell Carcinoma
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib will be administered orally at a dose of 60 mg/day continuously until 28 days prior to planned surgery or at time of the evidence of disease progression or onset of unacceptable toxicity.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib 60 mg/day orally
  Other Names: CABOMETYX

SUMMARY:
Cabozantinib in patients with advanced penile squamous cell carcinoma (PSCC): an open-label, single-center, phase 2, single-arm trial (CaboPen)

DETAILED DESCRIPTION:
an open-label, single-center, phase 2, single-arm trial

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Written informed consent
3. ECOG (Eastern Cooperative Oncology Group) performance status 0-1
4. Cytologically or histologically proven diagnosis of PSCC.
5. Histologically (Tru-cut biopsy) proven diagnosis of loco-regional nodal disease will be required in all cases except for those with clinical contraindications.
6. Uni- or bidimensionally measurable disease as defined by RECIST v1.1 criteria.
7. Clinical stage N2-3 and/or M1 (TNM 2002).
8. Locoregional relapse after prior major surgery/ies (either single or multiple).
9. No prior systemic therapy except for the administration of VBM (Vinblastine, Bleomycin, Methotrexate) chemotherapy for superficial disease if administered at least 6 months prior to study enrolment.
10. Adequate organ and marrow function .
11. Patients must be accessible for treatment and follow up as well as they must be willing and capable to comply with the requirements of the study. Patients registered on this trial must be treated and followed at the study sponsor site.

Exclusion Criteria:

1. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting.
   * Myocardial infarction.
   * Unstable angina.
   * Coronary artery by-pass graft surgery.
   * Symptomatic peripheral vascular disease.
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
   * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted during the study but should be used with caution - please refer to the study drug IB).
   * Screening ECG with a QTc>450 msec, congenital long QT syndrome, history of sustained ventricular tachycardia, history of ventricular fibrillation or torsade de pointes, bradycardia defined as heart rate < 50 bpm (patients with a pacemaker and heart rate > 50 bpm are eligible).
   * Uncontrolled hypertension.
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months ior to first dose of study drug.
3. History of HIV infection or active chronic hepatitis B or C.
4. Active clinically serious infections (> grade 2 NCI-CTC version 5.0).
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics).
6. Patients undergoing renal dialysis
7. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT treated basal cell carcinoma or any cancer curatively treated > 5 years prior to study entry.
8. History of clinically-significant gastrointestinal bleeding, inflammatory bowel disease, and other GI disorders associated with high risk of perforation or fistula formation or any other condition.
9. Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
10. Major surgery within 12 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment. Minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
11. History of allogenic organ solid transplantation.
12. Fertile males not willing to use a highly effective method of contraception or whose female partner is not using a highly effective contraception protection.
13. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
14. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.
15. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug.
16. Hemoptysis >=2.5 ml red blood within 3 months before treatment, signs indicative of pulmonary hemorrhage, cavitating pulmonary lesion, tumor invading major blood vessels and/or GI tract, endotracheal or endobronchial tumors History of clinically-significant gastrointestinal bleeding, inflammatory bowel disease, or any other condition among those listed in the full protocol.
17. Patients unable to swallow oral medications.
18. Concomitant anticoagulation with oral anticoagulants or platelet inhibitors.
19. History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
response -rate by RECIST v1.1 criteria | 40 months
  Assessment of response-rate by RECIST v1.1. Complete response + partial response

SECONDARY OUTCOMES:
Incidence of treatment-Emergent Adverse Event(safety and tolerability) | 40 months
  Assessment of the safety and tolerability: incidence, nature and severity of treatment-related adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Pathologic complete response (pCR) | 40 months
  Histological report of radical surgery
Progression-free survival (PFS). | 40 months
  Recist 1.1 criteria
Overall Survival (OS). | 40 months
  time will be calculated as the interval from treatment start date to the date of death for any cause, with censoring at the date of last contact for patients alive.
Variations of the Quality of Life | 40 months
  Variations of the Quality of Life score as assessed with the Edmonton Symptom Assessment Scale (ESAS), validated in Italian language. In this quality of life there are specify 9 main symptons: the score range is from 0 to 10 for each one.
  For each symptom the "0 score" corrisponds to "no symptom present" (better outcome) and the "10 score" corrisponds to "maximum symptom assessable" (worse outcome). The listed symptoms are: 1) Pain 2) Fatigue 3) Nausea 4) Depression 5) Anxiety 6) Somnolence 7) Loss of appetite 8) General Malaise 9) Dispnea. The total score is ranging from 0 to 90
FDG-PET/CT response rate according to EORTC criteria | 40 months
  1. to determine the rate of concordance with CT scan RECIST 1.1 response criteria and PET/CT EORTC Criteria
     * Complete response: complete disappearance of all target lesions with the exception of nodal disease (RECIST 1.1) and Complete resolution of FDG uptake in all lesions (EORTC)
     * Partial response (PR): greater than or equal to 30% decrease under baseline of the sum of target lesions (RECIST 1.1) and ≥ 25% reduction in the sum of SUVmax
     * Stable disease (SD): Not qualify for CR, PR or PD
     * Objective Progression (PD): 20% increase in the sum of diameters of target lesions or appearance of new unequivocal malignant lesions (RECIST 1.1) and ≥ 25% Increase in the sum of SUVmax or appearance of new lesions.
  2. To evaluate the relationship existing between tumor response measured by FDG-PET/CT EORTC Criteria (mainly early PET response as evaluated at first restaging) and pCR-rate (pT0 after surgery) and progression-free survival (months).

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Raggi, MD, Study Chair — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Barnholtz-Sloan JS, Maldonado JL, Pow-sang J, Giuliano AR. Incidence trends in primary malignant penile cancer. Urol Oncol. 2007 Sep-Oct;25(5):361-7. doi: 10.1016/j.urolonc.2006.08.029. PMID 17826651
- [Background] Ornellas AA. Management of penile cancer. J Surg Oncol. 2008 Mar 1;97(3):199-200. doi: 10.1002/jso.20893. No abstract available. PMID 17918225
- [Background] Misra S, Chaturvedi A, Misra NC. Penile carcinoma: a challenge for the developing world. Lancet Oncol. 2004 Apr;5(4):240-7. doi: 10.1016/S1470-2045(04)01427-5. PMID 15050955
- [Background] Heideman DA, Waterboer T, Pawlita M, Delis-van Diemen P, Nindl I, Leijte JA, Bonfrer JM, Horenblas S, Meijer CJ, Snijders PJ. Human papillomavirus-16 is the predominant type etiologically involved in penile squamous cell carcinoma. J Clin Oncol. 2007 Oct 10;25(29):4550-6. doi: 10.1200/JCO.2007.12.3182. PMID 17925550
- [Background] Li D, Han Z, Liu J, Zhang X, Ren J, Yan L, Liu H, Xu Z. Upregulation of nucleus HDGF predicts poor prognostic outcome in patients with penile squamous cell carcinoma bypass VEGF-A and Ki-67. Med Oncol. 2013 Dec;30(4):702. doi: 10.1007/s12032-013-0702-9. Epub 2013 Sep 3. PMID 23999841
- [Background] Zhu Y, Li H, Yao XD, Zhang SL, Zhang HL, Shi GH, Yang LF, Yang ZY, Wang CF, Ye DW. Feasibility and activity of sorafenib and sunitinib in advanced penile cancer: a preliminary report. Urol Int. 2010;85(3):334-40. doi: 10.1159/000315432. Epub 2010 Oct 27. PMID 20980789
- [Background] Bleeker MC, Heideman DA, Snijders PJ, Horenblas S, Dillner J, Meijer CJ. Penile cancer: epidemiology, pathogenesis and prevention. World J Urol. 2009 Apr;27(2):141-50. doi: 10.1007/s00345-008-0302-z. Epub 2008 Jul 8. PMID 18607597
- [Background] Bezerra AL, Lopes A, Santiago GH, Ribeiro KC, Latorre MR, Villa LL. Human papillomavirus as a prognostic factor in carcinoma of the penis: analysis of 82 patients treated with amputation and bilateral lymphadenectomy. Cancer. 2001 Jun 15;91(12):2315-21. PMID 11413520
- [Background] Backes DM, Kurman RJ, Pimenta JM, Smith JS. Systematic review of human papillomavirus prevalence in invasive penile cancer. Cancer Causes Control. 2009 May;20(4):449-57. doi: 10.1007/s10552-008-9276-9. Epub 2008 Dec 11. PMID 19082746
- [Background] Gregoire L, Cubilla AL, Reuter VE, Haas GP, Lancaster WD. Preferential association of human papillomavirus with high-grade histologic variants of penile-invasive squamous cell carcinoma. J Natl Cancer Inst. 1995 Nov 15;87(22):1705-9. doi: 10.1093/jnci/87.22.1705. PMID 7473819
- [Background] Miralles-Guri C, Bruni L, Cubilla AL, Castellsague X, Bosch FX, de Sanjose S. Human papillomavirus prevalence and type distribution in penile carcinoma. J Clin Pathol. 2009 Oct;62(10):870-8. doi: 10.1136/jcp.2008.063149. Epub 2009 Aug 25. PMID 19706632
- [Background] Rubin MA, Kleter B, Zhou M, Ayala G, Cubilla AL, Quint WG, Pirog EC. Detection and typing of human papillomavirus DNA in penile carcinoma: evidence for multiple independent pathways of penile carcinogenesis. Am J Pathol. 2001 Oct;159(4):1211-8. doi: 10.1016/S0002-9440(10)62506-0. PMID 11583947
- [Background] Mannweiler S, Sygulla S, Beham-Schmid C, Razmara Y, Pummer K, Regauer S. Penile carcinogenesis in a low-incidence area: a clinicopathologic and molecular analysis of 115 invasive carcinomas with special emphasis on chronic inflammatory skin diseases. Am J Surg Pathol. 2011 Jul;35(7):998-1006. doi: 10.1097/PAS.0b013e3182147e59. PMID 21681144
- [Background] Castellsague X, Bosch FX, Munoz N, Meijer CJ, Shah KV, de Sanjose S, Eluf-Neto J, Ngelangel CA, Chichareon S, Smith JS, Herrero R, Moreno V, Franceschi S; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Male circumcision, penile human papillomavirus infection, and cervical cancer in female partners. N Engl J Med. 2002 Apr 11;346(15):1105-12. doi: 10.1056/NEJMoa011688. PMID 11948269
- [Background] Backes DM, Bleeker MC, Meijer CJ, Hudgens MG, Agot K, Bailey RC, Ndinya-Achola JO, Hayombe J, Hogewoning CJ, Moses S, Snijders PJ, Smith JS. Male circumcision is associated with a lower prevalence of human papillomavirus-associated penile lesions among Kenyan men. Int J Cancer. 2012 Apr 15;130(8):1888-97. doi: 10.1002/ijc.26196. Epub 2011 Aug 2. PMID 21618520
- [Background] Barroso LF 2nd, Wilkin T. Human papillomavirus vaccination in males: the state of the science. Curr Infect Dis Rep. 2011 Apr;13(2):175-81. doi: 10.1007/s11908-010-0163-7. PMID 21365381
- [Background] Engels EA, Pfeiffer RM, Goedert JJ, Virgo P, McNeel TS, Scoppa SM, Biggar RJ; HIV/AIDS Cancer Match Study. Trends in cancer risk among people with AIDS in the United States 1980-2002. AIDS. 2006 Aug 1;20(12):1645-54. doi: 10.1097/01.aids.0000238411.75324.59. PMID 16868446
- [Background] Daling JR, Madeleine MM, Johnson LG, Schwartz SM, Shera KA, Wurscher MA, Carter JJ, Porter PL, Galloway DA, McDougall JK, Krieger JN. Penile cancer: importance of circumcision, human papillomavirus and smoking in in situ and invasive disease. Int J Cancer. 2005 Sep 10;116(4):606-16. doi: 10.1002/ijc.21009. PMID 15825185
- [Background] Hellberg D, Valentin J, Eklund T, Nilsson S. Penile cancer: is there an epidemiological role for smoking and sexual behaviour? Br Med J (Clin Res Ed). 1987 Nov 21;295(6609):1306-8. doi: 10.1136/bmj.295.6609.1306. PMID 3120988
- [Background] Marconnet L, Rigaud J, Bouchot O. Long-term followup of penile carcinoma with high risk for lymph node invasion treated with inguinal lymphadenectomy. J Urol. 2010 Jun;183(6):2227-32. doi: 10.1016/j.juro.2010.02.025. PMID 20399455
- [Background] Protzel C, Alcaraz A, Horenblas S, Pizzocaro G, Zlotta A, Hakenberg OW. Lymphadenectomy in the surgical management of penile cancer. Eur Urol. 2009 May;55(5):1075-88. doi: 10.1016/j.eururo.2009.02.021. Epub 2009 Feb 23. PMID 19264390
- [Background] Heyns CF, Fleshner N, Sangar V, Schlenker B, Yuvaraja TB, van Poppel H. Management of the lymph nodes in penile cancer. Urology. 2010 Aug;76(2 Suppl 1):S43-57. doi: 10.1016/j.urology.2010.03.001. PMID 20691885
- [Background] Pompeo AC. Extended lymphadenectomy in penile cancer. Can J Urol. 2005 Feb;12 Suppl 1:30-6; discussion 97-8. PMID 15780162
- [Background] Kroon BK, Horenblas S, Lont AP, Tanis PJ, Gallee MP, Nieweg OE. Patients with penile carcinoma benefit from immediate resection of clinically occult lymph node metastases. J Urol. 2005 Mar;173(3):816-9. doi: 10.1097/01.ju.0000154565.37397.4d. PMID 15711276
- [Background] Lont AP, Kroon BK, Gallee MP, van Tinteren H, Moonen LM, Horenblas S. Pelvic lymph node dissection for penile carcinoma: extent of inguinal lymph node involvement as an indicator for pelvic lymph node involvement and survival. J Urol. 2007 Mar;177(3):947-52; discussion 952. doi: 10.1016/j.juro.2006.10.060. PMID 17296384
- [Background] Ornellas AA, Kinchin EW, Nobrega BL, Wisnescky A, Koifman N, Quirino R. Surgical treatment of invasive squamous cell carcinoma of the penis: Brazilian National Cancer Institute long-term experience. J Surg Oncol. 2008 May 1;97(6):487-95. doi: 10.1002/jso.20980. PMID 18425779
- [Background] Spiess PE, Izawa JI, Bassett R, Kedar D, Busby JE, Wong F, Eddings T, Tamboli P, Pettaway CA. Preoperative lymphoscintigraphy and dynamic sentinel node biopsy for staging penile cancer: results with pathological correlation. J Urol. 2007 Jun;177(6):2157-61. doi: 10.1016/j.juro.2007.01.125. PMID 17509308
- [Background] Izawa J, Kedar D, Wong F, Pettaway CA. Sentinel lymph node biopsy in penile cancer: evolution and insights. Can J Urol. 2005 Feb;12 Suppl 1:24-9. PMID 15780161
- [Background] Hungerhuber E, Schlenker B, Frimberger D, Linke R, Karl A, Stief CG, Schneede P. Lymphoscintigraphy in penile cancer: limited value of sentinel node biopsy in patients with clinically suspicious lymph nodes. World J Urol. 2006 Aug;24(3):319-24. doi: 10.1007/s00345-006-0073-3. Epub 2006 Apr 11. PMID 16688459
- [Background] Neto AS, Tobias-Machado M, Ficarra V, Wroclawski ML, Amarante RD, Pompeo AC, Del Giglio A. Dynamic sentinel node biopsy for inguinal lymph node staging in patients with penile cancer: a systematic review and cumulative analysis of the literature. Ann Surg Oncol. 2011 Jul;18(7):2026-34. doi: 10.1245/s10434-010-1546-6. Epub 2011 Feb 10. PMID 21308487
- [Background] Graafland NM, Valdes Olmos RA, Meinhardt W, Bex A, van der Poel HG, van Boven HH, Nieweg OE, Horenblas S. Nodal staging in penile carcinoma by dynamic sentinel node biopsy after previous therapeutic primary tumour resection. Eur Urol. 2010 Nov;58(5):748-51. doi: 10.1016/j.eururo.2010.06.036. Epub 2010 Jul 12. PMID 20633981
- [Background] Pettaway CA, Pisters LL, Dinney CP, Jularbal F, Swanson DA, von Eschenbach AC, Ayala A. Sentinel lymph node dissection for penile carcinoma: the M. D. Anderson Cancer Center experience. J Urol. 1995 Dec;154(6):1999-2003. PMID 7500444
- [Background] Pizzocaro G, Algaba F, Horenblas S, Solsona E, Tana S, Van Der Poel H, Watkin NA; European Association of Urology (EAU) Guidelines Group on Penile Cancer. EAU penile cancer guidelines 2009. Eur Urol. 2010 Jun;57(6):1002-12. doi: 10.1016/j.eururo.2010.01.039. Epub 2010 Feb 4. PMID 20163910
- [Background] Gagliano RG, Blumenstein BA, Crawford ED, Stephens RL, Coltman CA Jr, Costanzi JJ. cis-Diamminedichloroplatinum in the treatment of advanced epidermoid carcinoma of the penis: a Southwest Oncology Group Study. J Urol. 1989 Jan;141(1):66-7. doi: 10.1016/s0022-5347(17)40590-8. PMID 2642312
- [Background] Leijte JA, Kirrander P, Antonini N, Windahl T, Horenblas S. Recurrence patterns of squamous cell carcinoma of the penis: recommendations for follow-up based on a two-centre analysis of 700 patients. Eur Urol. 2008 Jul;54(1):161-8. doi: 10.1016/j.eururo.2008.04.016. Epub 2008 Apr 15. PMID 18440124
- [Background] Culkin DJ, Beer TM. Advanced penile carcinoma. J Urol. 2003 Aug;170(2 Pt 1):359-65. doi: 10.1097/01.ju.0000062829.43654.5e. PMID 12853775
- [Background] Pizzocaro G, Piva L. Adjuvant and neoadjuvant vincristine, bleomycin, and methotrexate for inguinal metastases from squamous cell carcinoma of the penis. Acta Oncol. 1988;27(6b):823-4. doi: 10.3109/02841868809094366. PMID 2466471
- [Background] Leijte JA, Kerst JM, Bais E, Antonini N, Horenblas S. Neoadjuvant chemotherapy in advanced penile carcinoma. Eur Urol. 2007 Aug;52(2):488-94. doi: 10.1016/j.eururo.2007.02.006. Epub 2007 Feb 14. PMID 17316964
- [Background] Hakenberg OW, Nippgen JB, Froehner M, Zastrow S, Wirth MP. Cisplatin, methotrexate and bleomycin for treating advanced penile carcinoma. BJU Int. 2006 Dec;98(6):1225-7. doi: 10.1111/j.1464-410X.2006.06496.x. PMID 17125480
- [Background] Bermejo C, Busby JE, Spiess PE, Heller L, Pagliaro LC, Pettaway CA. Neoadjuvant chemotherapy followed by aggressive surgical consolidation for metastatic penile squamous cell carcinoma. J Urol. 2007 Apr;177(4):1335-8. doi: 10.1016/j.juro.2006.11.038. PMID 17382727
- [Background] Pagliaro LC, Williams DL, Daliani D, Williams MB, Osai W, Kincaid M, Wen S, Thall PF, Pettaway CA. Neoadjuvant paclitaxel, ifosfamide, and cisplatin chemotherapy for metastatic penile cancer: a phase II study. J Clin Oncol. 2010 Aug 20;28(24):3851-7. doi: 10.1200/JCO.2010.29.5477. Epub 2010 Jul 12. PMID 20625118
- [Background] Graafland NM, Valdes Olmos RA, Teertstra HJ, Kerst JM, Bergman AM, Horenblas S. 18F-FDG PET/CT for monitoring induction chemotherapy in patients with primary inoperable penile carcinoma: first clinical results. Eur J Nucl Med Mol Imaging. 2010 Aug;37(8):1474-80. doi: 10.1007/s00259-010-1434-0. Epub 2010 Mar 27. PMID 20349185
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Hitt R, Lopez-Pousa A, Martinez-Trufero J, Escrig V, Carles J, Rizo A, Isla D, Vega ME, Marti JL, Lobo F, Pastor P, Valenti V, Belon J, Sanchez MA, Chaib C, Pallares C, Anton A, Cervantes A, Paz-Ares L, Cortes-Funes H. Phase III study comparing cisplatin plus fluorouracil to paclitaxel, cisplatin, and fluorouracil induction chemotherapy followed by chemoradiotherapy in locally advanced head and neck cancer. J Clin Oncol. 2005 Dec 1;23(34):8636-45. doi: 10.1200/JCO.2004.00.1990. Epub 2005 Nov 7. PMID 16275937
- [Background] Maiche AG. Adjuvant treatment using bleomycin in squamous cell carcinoma of penis: study of 19 cases. Br J Urol. 1983 Oct;55(5):542-4. doi: 10.1111/j.1464-410x.1983.tb03366.x. PMID 6194844
- [Background] Protzel C, Ruppin S, Milerski S, Klebingat KJ, Hakenberg OW. [The current state of the art of chemotherapy of penile cancer: results of a nationwide survey of German clinics]. Urologe A. 2009 Dec;48(12):1495-8. doi: 10.1007/s00120-009-2108-z. German. PMID 19774356
- [Background] Corral DA, Sella A, Pettaway CA, Amato RJ, Jones DM, Ellerhorst J. Combination chemotherapy for metastatic or locally advanced genitourinary squamous cell carcinoma: a phase II study of methotrexate, cisplatin and bleomycin. J Urol. 1998 Nov;160(5):1770-4. PMID 9783949
- [Background] Dexeus FH, Logothetis CJ, Sella A, Amato R, Kilbourn R, Fitz K, Striegel A. Combination chemotherapy with methotrexate, bleomycin and cisplatin for advanced squamous cell carcinoma of the male genital tract. J Urol. 1991 Nov;146(5):1284-7. doi: 10.1016/s0022-5347(17)38069-2. PMID 1719241
- [Background] Haas GP, Blumenstein BA, Gagliano RG, Russell CA, Rivkin SE, Culkin DJ, Wolf M, Crawford ED. Cisplatin, methotrexate and bleomycin for the treatment of carcinoma of the penis: a Southwest Oncology Group study. J Urol. 1999 Jun;161(6):1823-5. PMID 10332445
- [Background] Pettaway CA, Pagliaro L, Theodore C, Haas G. Treatment of visceral, unresectable, or bulky/unresectable regional metastases of penile cancer. Urology. 2010 Aug;76(2 Suppl 1):S58-65. doi: 10.1016/j.urology.2010.03.082. PMID 20691886
- [Background] Pizzocaro G, Nicolai N, Milani A. Taxanes in combination with cisplatin and fluorouracil for advanced penile cancer: preliminary results. Eur Urol. 2009 Mar;55(3):546-51. doi: 10.1016/j.eururo.2008.07.014. Epub 2008 Jul 14. PMID 18649992
- [Background] Trabulsi EJ, Hoffman-Censits J. Chemotherapy for penile and urethral carcinoma. Urol Clin North Am. 2010 Aug;37(3):467-74. doi: 10.1016/j.ucl.2010.04.010. PMID 20674701
- [Background] Hussein AM, Benedetto P, Sridhar KS. Chemotherapy with cisplatin and 5-fluorouracil for penile and urethral squamous cell carcinomas. Cancer. 1990 Feb 1;65(3):433-8. doi: 10.1002/1097-0142(19900201)65:33.0.co;2-g. PMID 2297633
- [Background] Shammas FV, Ous S, Fossa SD. Cisplatin and 5-fluorouracil in advanced cancer of the penis. J Urol. 1992 Mar;147(3):630-2. doi: 10.1016/s0022-5347(17)37327-5. PMID 1538445
- [Background] Di Lorenzo G, Buonerba C, Federico P, Perdona S, Aieta M, Rescigno P, D'Aniello C, Puglia L, Petremolo A, Ferro M, Marinelli A, Palmieri G, Sonpavde G, Mirone V, De Placido S. Cisplatin and 5-fluorouracil in inoperable, stage IV squamous cell carcinoma of the penis. BJU Int. 2012 Dec;110(11 Pt B):E661-6. doi: 10.1111/j.1464-410X.2012.11453.x. Epub 2012 Sep 10. PMID 22958571
- [Background] Theodore C, Skoneczna I, Bodrogi I, Leahy M, Kerst JM, Collette L, Ven K, Marreaud S, Oliver RDT; EORTC Genito-Urinary Tract Cancer Group. A phase II multicentre study of irinotecan (CPT 11) in combination with cisplatin (CDDP) in metastatic or locally advanced penile carcinoma (EORTC PROTOCOL 30992). Ann Oncol. 2008 Jul;19(7):1304-1307. doi: 10.1093/annonc/mdn149. Epub 2008 Apr 15. PMID 18417462
- [Background] Power DG, Galvin DJ, Cuffe S, McVey GP, Mulholland PJ, Farrelly C, Delaney DW, O'Byrne KJ. Cisplatin and gemcitabine in the management of metastatic penile cancer. Urol Oncol. 2009 Mar-Apr;27(2):187-90. doi: 10.1016/j.urolonc.2007.10.015. Epub 2008 Feb 4. PMID 18367122
- [Background] Di Lorenzo G, Federico P, Buonerba C, Longo N, Carteni G, Autorino R, Perdona S, Ferro M, Rescigno P, D'Aniello C, Matano E, Altieri V, Palmieri G, Imbimbo C, De Placido S, Mirone V. Paclitaxel in pretreated metastatic penile cancer: final results of a phase 2 study. Eur Urol. 2011 Dec;60(6):1280-4. doi: 10.1016/j.eururo.2011.08.028. Epub 2011 Aug 22. PMID 21871710
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Moro C, Brunelli C, Miccinesi G, Fallai M, Morino P, Piazza M, Labianca R, Ripamonti C. Edmonton symptom assessment scale: Italian validation in two palliative care settings. Support Care Cancer. 2006 Jan;14(1):30-7. doi: 10.1007/s00520-005-0834-3. Epub 2005 Jun 4. PMID 15937688
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991